CLINICAL TRIAL: NCT02028819
Title: Compassionate Use of Ibalizumab for the Treatment of HIV Infection
Status: No longer available | Type: Expanded Access
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0003
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; ibalizumab

INTERVENTIONS:
Drug: Dolutegravir Sodium Monohydrate — Dolutegravir taken 50mg orally twice daily
  Other Names: TIVICAY
Drug: Ibalizumab — Ibalizumab will be administered intravenously at a dose of 800mg once every two weeks.
  Other Names: TMB-355

SUMMARY:
Ibalizumab is a humanized immunoglobulin G monoclonal antibody directed against a human T-cell receptor (CD4) and thus suppresses HIV replication by blocking entry of HIV into CD4+ lymphocytes. Ibalizumab has completed phase I and II clinical studies in HIV-negative and HIV-infected individuals showing safety and efficacy for suppressing HIV replication.

DETAILED DESCRIPTION:
1. Ibalizumab is a humanized immunoglobulin G monoclonal antibody directed against a human T-cell receptor (CD4) and thus suppresses HIV replication by blocking entry of HIV into CD4+ lymphocytes. Ibalizumab is in the pipeline for FDA approval to treat HIV infection. Phase I and II clinical studies have been completed in HIV-negative and HIV-infected individuals showing safety and efficacy for suppressing HIV replication.
2. Use of this medication requires that a single patient IND be obtained from the FDA for each patient requiring ibalizumab. An individual use IND has been approved by the FDA for one patient on treatment through this protocol; The IND number is 114515. The manufacturer of ibalizumab (TaiMed Biologics, Inc) will ship the drug directly to the Denver Health pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of HIV-infection with resistance or intolerance to currently available antiretroviral medications available in the United States or in whom additional drugs need to be added to their regimen because of inadequate response to existing therapy
* Patients with HIV infection that is expected to be sensitive to dolutegravir and ibalizumab
* Patients who do not qualify for or who are otherwise ineligible for clinical trials of medications not currently approved for treatment of HIV infection in the U.S.

Exclusion Criteria:

* Patients who are allergic to or have had a severe adverse reaction to dolutegravir or ibalizumab in the past.
* Age <18 years or >89 years
* Women may not be pregnant
* Prisoners and decisionally challenged patients will be excluded

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Gardner, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Health, Denver, Colorado, United States